CLINICAL TRIAL: NCT00006433
Title: Phase I/II Trial of Doxil and Hyperthermia for Breast Cancer Patients With Chest Wall Recurrence or Stage IV Disease With Locally Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Purpose: Treatment
Other Study IDs: NCRR-M01RR00030-0156; M01RR000030 (NIH)
Record Dates: First submitted 2000-11-03; First posted 2000-11-06 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Diathermy

INTERVENTIONS:
Drug: Doxil
Procedure: heat treatment

SUMMARY:
Purpose: The purpose of this protocol is to evaluate the combination of Doxil chemotherapy and heat treatment for recurrent breast cancer located on the chestwall following mastectomy. This protocol also includes patients with metastatic breast cancer who have not had mastectomy but have advanced tumor remaining within the breast. Doxil is the drug adriamycin (also called doxorubicin) encapsulated in liposomes, which coats the drug with a small amount of lipid (fat). This chemotherapy is in a newer form which can be better delivered to the tumor tissue without causing as much systemic toxicity. We are combining heat treatment with this drug in an effort to further increase the delivery of drug to the tumor, which may give an increased tumor response.

Methods: The patients will be treated with chemotherapy followed by heat treatment. This will be given for 6 cycles approximately every 4 weeks. For the first cycle patients will need to be hospitalized 3 days for measurement of blood levels of drug as well as some additional radiology studies which will help us to determine whether the drug is preferentially distributed within tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent or metastatic breast cancer

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01

CONTACTS AND LOCATIONS:
Overall Officials: Leonard R. Prosnitz, M.D., Principal Investigator
Locations (1):
- Radiation Oncology, Duke University Medical Center, Durham, North Carolina, United States